CLINICAL TRIAL: NCT02039570
Title: Investigating the Relationship Between Haemorrhoids, Internal Iliac Veins and Tributary Reflux
Brief Title: The Relationship Between Haemorrhoids and Pelvic Vein Reflux
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: HaemorrhoidsJan2104
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Haemorrhoids
Keywords: haemorrhoids; pelvic reflux
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- haemorrhoids: The cohort contains only patients with symptomatic haemorrhoids - these patients will receive a transvaginal scan to examine their ovarian and internal iliac veins to ascertain whether there is any reflux
  Interventions: Other: Transvaginal scan

INTERVENTIONS:
Other: Transvaginal scan — transvaginal scan conducted using duplex ultrasonography

SUMMARY:
This case series aims to find out in a group of female patients suffering from haemorrhoids, how many of them have pelvic vein reflux that feeds into their haemorrhoids.

This will be done by examining their ovarian and internal iliac veins for reflux, using a transvaginal scan.

DETAILED DESCRIPTION:
Based on previous research, we believe that haemorrhoids could be caused by faulty valves in the veins running from deep within the pelvic region to the lower part of the abdomen (internal iliac veins)resulting in reflux in the tributaries.

We have already presented research showing that patients with severe pelvic vein reflux, particularly of the internal iliac veins and tributaries, are associated with a higher chance of haemorrhoids.

The aim of this study is to see in a group of patients suffering from haemorrhoids, whether all of them exhibit pelvic vein reflux feeding into the haemorrhoids.

If we are able to prove that either all or the vast majority of patients with true haemorrhoids do have pelvic vein reflux feeding into them, this will support our hypothesis that the internal iliac vein and tributary reflux is causative of haemorrhoids.

following this, in a future study we will treat internal iliac vein and tributary reflux to see if the results of haemorrhoid treatments are improved.

If we find only a few patients with haemorrhoids have associated internal iliac vein and tributary reflux feeding into the haemorrhoids, we will be able to refute the hypothesis that there is a causative association, and will not need to progress with the studies and will look instead for a different aetiology.

At the current time, there is no effective way of investigating male pelvic vein reflux. The gold standard investigation for pelvic vein reflux is transvaginal duplex ultrasound scan. As such this study will be restricted to females presenting with symptomatically haemorrhoids who are able and willing to undergo transvaginal ultrasound scan to assess their pelvic veins.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Symptomatic haemorrhoids
* Being able and willing to undergo transvaginal ultrasound scan to assess their ovarian and internal iliac veins
* Aged between 18 and 80 years
* good understanding of written and spoken english

Exclusion Criteria:

* male
* aged younger than 18 or older than 80
* Those unwilling to attend for a transvaginal scan at The Whiteley Clinic, Guildford

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the sample will be selected from female patients presenting in primary care with symptomatic haemorrhoids
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Reflux in ovarian veins | Immediatley
  Following a transvaginal scan pelvic reflux in both the right and left leg separately will be rated on a four point scale 0 no reflux
  1. trickle reflux
  2. significant reflux
  3. severe reflux

OTHER OUTCOMES:
Reflux in internal iliac veins | immediatley
  internal iliac veins in the left and right legs will be rated using the following scale 0 no reflux
  1. trickle reflux
  2. significant reflux
  3. severe reflux
Goligher classification | immedialtey
  The Goligher classification will be used to rate the severity of the participants' haemorrhoids

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteley, Professor, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Surrey, Guildford, United Kingdom